CLINICAL TRIAL: NCT03412396
Title: A Single Arm Study of 6-Months Neoadjuvant Apalutamide Prior to Radical Prostatectomy in Intermediate Risk Patients to Reduce the Frequency of Pathologic Features That Drive Post-Operative Radiation Therapy
Brief Title: Apalutamide in Treating Patients With Prostate Cancer Before Radical Prostatectomy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0693; NCI-2018-00902 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0693 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Prostate Adenocarcinoma; Stage IIB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (apalutamide, radical prostatectomy) (Experimental): Patients receive apalutamide PO daily for 24 weeks in the absence of disease progression or unacceptable toxicity. Within 2 weeks of completing apalutamide, patients undergo radical prostatectomy.
  Interventions: Drug: Apalutamide; Other: Quality-of-Life Assessment; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Radical Prostatectomy — Undergo radical prostatectomy
  Other Names: Prostatovesiculectomy

SUMMARY:
This phase II trial studies how well apalutamide works in treating patients with prostate cancer before radical prostatectomy. Androgen can cause the growth of prostate cancer cells. Hormone therapy using apalutamide may fight prostate cancer by lowering the amount of androgen the body makes and may make it less likely for patients to receive radiation therapy after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether 6 months (24 weeks) of neoadjuvant apalutamide prior to prostatectomy for intermediate risk prostate cancer results in a reduction of aggregate pathologic risk features that drive post-operative radiotherapy recommendations from 35% to 15%.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of 6 months (24 weeks) neoadjuvant apalutamide followed by radical prostatectomy for intermediate risk prostate cancer.

II. To estimate the frequency of clinical complete responses and "near" complete responses (currently defined as < 6 mm total tumor volume).

III. To characterize the molecular features of the treated prostate cancers and link them to morphologic characterization.

IV. To measure the 3-5 year biochemical recurrence rate of treated patients as a baseline to inform a larger phase III trial.

OUTLINE:

Patients receive apalutamide orally (PO) daily for 24 weeks in the absence of disease progression or unacceptable toxicity. Within 2 weeks of completing apalutamide, patients undergo radical prostatectomy.

After completion of study treatment, patients are followed up at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Histologically confirmed adenocarcinoma of the prostate
* A minimum of 10 core biopsies have been performed at baseline and available. A prostate biopsy within 6 months from screening is allowed for entry requirements. Biopsies performed within 6-12 months from screening are acceptable if the treating physician would allow treatment without further biopsy. Patients must meet intermediate risk criteria from Gleason score, T stage, and prostate-specific antigen (PSA) value by National Comprehensive Cancer Network (NCCN) criteria: cT2b-T2c or Gleason 7 (3+4 or 4+3) or PSA 10-20 ng/mL. In addition, the Gleason 3+4 or 4+3 must be present
* Pathology review at MD Anderson Cancer Center. The volume of disease must be high enough for the surgeon to agree to include an extended template pelvic lymph node dissection
* Serum testosterone > 200 ng/mL
* Patient and urologist must agree that patient is suitable for prostatectomy
* No evidence of metastases on imaging. This risk group does not require metastatic studies, but if performed they must be negative (as determined by urologist or radiologist). Suspicious lymph nodes permissible if < 10 mm
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Hemoglobin >= 10.0 g/dL
* Platelet count >= 100,000 x 10^9/microliter
* Glomerular filtration rate (GFR) >= 45 mL/min
* Serum potassium >= 3.5 mmol/L
* Serum albumin >= 3.0 g/dL
* Able to swallow the study drug whole as a tablet
* Serum bilirubin < 1.5 x upper limit of normal (ULN); Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject may be eligible
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN
* Normal coagulation profile and no history of substantial non-iatrogenic bleeding diathesis
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Histological variants in the primary tumor, other than adenocarcinoma; for example: neuroendocrine tumor, small cell or sarcomatoid
* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* PSA is > than 20 ng/mL (NOTE: unless other valid PSAs were =< 20 and the treating physician considers a value > 20 related to the biopsy or other non-malignant cause. The treating physician must consider the patient intermediate risk in aggregate)
* Uncontrolled hypertension. Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy. Note that this is NOT a criterion related to particular blood pressure (BP) results at the time of assessment for eligibility, nor does it apply to acute BP excursions that are related to iatrogenic causes, acute pain or other transient, reversible causes
* Active or symptomatic viral hepatitis or chronic liver disease
* Clinically significant heart disease as evidenced by myocardial infarction, arterial thrombotic events in the past 6 months, severe or unstable angina, class III-IV New York Heart Association heart failure
* Other malignancy, except non-melanoma skin cancer, that is active or has a >= 30% probability of recurrence within 12 months
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug
* Known history of pituitary and/or adrenal disease (or dysfunction)
* Prior hormone therapy for prostate cancer including orchiectomy, antiandrogens, ketoconazole, or estrogens (5-alpha reductase inhibitors allowed), or luteinizing hormone-releasing hormone (LHRH) agonists/antagonists
* Severely compromised immunological state, including being positive for the human immunodeficiency virus (HIV)
* Patients who are not appropriate surgical candidates for radical prostatectomy based on the evaluation of co-existent medical diseases and competing potential causes of death (such as but not limited to, unstable angina, myocardial infarction within the previous 6 months, or use of ongoing maintenance therapy for life-threatening ventricular arrhythmia, uncontrolled hypertension)
* History of seizure, seizure disorder, or any condition that may predispose to seizure including, but not limited to underlying brain injury, stroke, primary brain tumors, brain metastases, or alcoholism. Also, history of loss of consciousness or transient ischemic attack within 12 months of enrollment (day 1 visit). Drugs may not be used which are known to decrease the seizure threshold

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2026-03-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John W Davis, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2018 and February 2020, 45 men were enrolled, initiated preoperative apalutamide, and were evaluable for safety outcomes. Of those, two patients withdrew consent prior to surgery, one patient stopped apalutamide at <9 weeks after initiation, and two patients did not undergo a Radical Prostatectomy (RP)
Groups:
- Open label apalutamide and surgery: apalutamide 240 mg/day orally for a total duration of 24 weeks, and RP plus ePLND was performed within 3 weeks of completing apalutamide
Period: Overall Study
Arm/Group | Open label apalutamide and surgery
Started | 45
Completed | 40
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — "stopped apalutamide at <9 weeks after initiation" | 1
Not completed — Did not undergo RP | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open label apalutamide and surgery
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 60 [56.8 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Surgical Pathology Features at Risk of Pelvic Radiation Therapy
Description: To determine whether 6 months (24 weeks) of neoadjuvant apalutamide prior to prostatectomy for intermediate risk prostate cancer results in a reduction of surgical pathology features at risk of pelvic RT, defined as pT3a, pT3b stage, N1 and/or positive surgical margin. All patients who receive at least 9 weeks of neoadjuvant therapy of apalutamide and undergo radical prostatectomy will be evaluable for the primary endpoint.
Time Frame: Assessed at time of surgical specimen microscopic evalution Assessed at time of surgical specimen microscopic evaluation
Measure: Count of Participants; unit: Participants
Groups:
- Open label apalutamide and surgery: apalutamide 240 mg/day orally for a total duration of 24 weeks, and RP (radical prostatectomy) plus ePLND was performed within 3 weeks of completing apalutamide
Arm/Group | Open label apalutamide and surgery
Number analyzed (Participants) | 40
Participants | 16

2. Secondary Outcome: Safety and Tolerability of 6 Months Neoadjuvant Apalutamide Followed by Radical Prostatectomy
Description: Incidence of treatment emergent adverse events (TEAEs). All patients who receive any dose of apalutamide will be evaluable for safety.
Time Frame: From initiation of apalutamide through 30 days post-surgery. For those participants who did not have surgery, we assessed the reported AEs until 30 days after the last dose of apalutamide.
Measure: Count of Participants; unit: Participants
Arm/Group | Open label apalutamide and surgery
Number analyzed (Participants) | 45
Participants
  Any TEAEs | 45
  Grade ≥3 TEAE | 13
  TEAE leading to discontinuation | 4

3. Secondary Outcome: Clinical Complete Responses (pT0) and "Near" Complete Responses (<6mm Total Tumor Volume)
Description: The numbers of patients with <6 mm total tumor volume in their surgical specimens, assessed by study Pathologist.
Time Frame: Assessed at time of surgical specimen microscopic evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Open label apalutamide and surgery
Number analyzed (Participants) | 40
Participants | 0

4. Secondary Outcome: Biochemical Recurrence Rate
Description: Number of patients who had a PSA value of equal of more than 0.2 ng/dL after surgery and through 3 years of follow up.
Time Frame: From surgery through 3-year post-op follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Open label apalutamide and surgery
Number analyzed (Participants) | 40
Participants | 6

ADVERSE EVENTS:
Time Frame: From initiation of apalutamide through 30 days post-surgery. For those participants who did not have surgery, we assessed the reported AEs until 30 days after the last dose of apalutamide.
Arm/Group | Open label apalutamide and surgery
All-Cause Mortality (participants affected / at risk) | 1/45
Serious Adverse Events (participants affected / at risk) | 2/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open label apalutamide and surgery (N=45)
Death NOS (Cardiac disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open label apalutamide and surgery (N=45)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 10 (10)
Anemia (Blood and lymphatic system disorders) | 15 (15)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10)
AST elevated (Blood and lymphatic system disorders) | 5 (5)
ALT elevated (Blood and lymphatic system disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (5)
Creatinine elevated (Blood and lymphatic system disorders) | 5 (5)
Decreased libido (General Disorders) | 9 (9)
Depression (General Disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 6 (6)
Dysgeusia (Gastrointestinal disorders) | 5 (5)
Edema (Blood and lymphatic system disorders) | 3 (3)
Elevated TSH (Blood and lymphatic system disorders) | 10 (10)
Elevated testosterone (Blood and lymphatic system disorders) | 20 (20)
Fatigue (General disorders) | 17 (19)
Gynecomastia (Reproductive system and breast disorders) | 20 (20)
Erectile Dysfunction (Reproductive system and breast disorders) | 10 (10)
Headache (Nervous system disorders) | 5 (5)
Hypertension (Nervous system disorders) | 6 (7)
Hypophosphatemia (Blood and lymphatic system disorders) | 6 (6)
Insomnia (Nervous system disorders) | 8 (8)
Hyperglycemia (Blood and lymphatic system disorders) | 11 (12)
Weight loss (Metabolism and nutrition disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03412396/Prot_SAP_000.pdf